CLINICAL TRIAL: NCT00558844
Title: Phase 1b/2a Multidose Safety and Tolerability Study of Liposomal Amikacin for Inhalation (Arikayce™) in Cystic Fibrosis Patient With Chronic Infections Due to Pseudomonas Aeruginosa.
Brief Title: Safety/Tolerability Study of Arikayce™ in Cystic Fibrosis Patients With Chronic Infection Due to Pseudomonas Aeruginosa
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Insmed Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TR02-106
Record Dates: First submitted 2007-11-13; First posted 2007-11-15 (Estimated); Results first posted 2019-06-04 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Respiratory Infections; Pulmonary Cystic Fibrosis; CFTR
MeSH Terms: conditions — Cystic Fibrosis; Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- A (Active Comparator): Arikayce™ at 560 mg Subjects randomized 2:1 to receive Arikayce 560 mg or Placebo.
  Interventions: Drug: Arikayce™ 560 mg
- B (Placebo Comparator): Matching placebo for 560 mg Subjects randomized 2:1 to receive Arikayce 560 mg or Placebo.
  Interventions: Drug: Placebo for 560 mg
- C (Active Comparator): Arikayce™ at 70 mg Subjects randomized 1:1:1 to receive Arikayce 70 mg, Arikayce 140 mg or Placebo.
  Interventions: Drug: Arikayce™ 70 mg
- D (Active Comparator): Arikayce™ at 140 mg Subjects randomized 1:1:1 to receive Arikayce 70 mg, Arikayce 140 mg or Placebo.
  Interventions: Drug: Arikayce™ 140 mg
- E (Placebo Comparator): Matching placebo for 70 mg/140 mg Subjects randomized 1:1:1 to receive Arikayce 70 mg, Arikayce 140 mg or Placebo.
  Interventions: Drug: Placebo for 70 mg / 140 mg

INTERVENTIONS:
Drug: Arikayce™ 560 mg — Arikayce™ at 560 mg
  Subjects will be randomly assigned to study drug dose of of Arikayce™ or placebo in accordance with a code provided by the Sponsor/CRO. Randomization will be made in a 2:1 allocation between Arikayce™ and placebo. They will be blinded whether they receive Arikayce™ or Placebo Study subjects will receive Arikayce™ or placebo on Days 1 through Day 28. Drug is administered once a day via a nebulizer.
  Arms: A
Drug: Placebo for 560 mg — Matching placebo
  Subjects will be randomly assigned to study drug dose of of Arikayce™ or placebo in accordance with a code provided by the Sponsor/CRO. Randomization will be made in a 2:1 allocation between Arikayce™ and placebo. They will be blinded whether they receive Arikayce™ or Placebo Study subjects will receive Arikayce™ or placebo on Days 1 through Day 28. Drug is administered once a day via a nebulizer.
  Arms: B
Drug: Arikayce™ 70 mg — Subjects will be randomly assigned to study drug dose of of Arikayce™ or placebo in accordance with a code provided by the Sponsor/CRO. Randomization will be made in a 1:1:1 allocation between Arikayce™ and placebo. They will be blinded whether they receive Arikayce™ or Placebo Study subjects will receive Arikayce™ or placebo on Days 1 through Day 28. Drug is administered once a day via a nebulizer.
  Arms: C
Drug: Arikayce™ 140 mg — Subjects will be randomly assigned to study drug dose of of Arikayce™ or placebo in accordance with a code provided by the Sponsor/CRO. Randomization will be made in a 1:1:1 allocation between Arikayce™ and placebo. They will be blinded whether they receive Arikayce™ or Placebo Study subjects will receive Arikayce™ or placebo on Days 1 through Day 28. Drug is administered once a day via a nebulizer.
  Arms: D
Drug: Placebo for 70 mg / 140 mg — Matching placebo
  Subjects will be randomly assigned to study drug dose of of Arikayce™ or placebo in accordance with a code provided by the Sponsor/CRO. Randomization will be made in a 1:1:1 allocation between Arikayce™ and placebo. They will be blinded whether they receive Arikayce™ or Placebo Study subjects will receive Arikayce™ or placebo on Days 1 through Day 28. Drug is administered once a day via a nebulizer.
  Arms: E

SUMMARY:
This is a study to determine the safety and tolerability of 28 days of daily dosing of 560 mg of Arikayce™ versus placebo and daily dosing of 70 mg and 140 mg of Arikayce™ versus placebo in patients who have Cystic fibrosis (CF) and chronic infection due to pseudomonas aeruginosa.

DETAILED DESCRIPTION:
CF is a gentic disease resulting from mutations in a 230 kb gene on chromosome 7 known as the cystic fibrosis transmembrane conductance regulator (CFTR). Study subjects with CF manifest pathological changes in a variety or organs that express CFTR. The lungs are frequently affected, the sequelae being chronic infections and airway inflammation. The principal goal of both treatment of subjects with CF is to slow the chronic deterioration of lung function.

Study subjects will be randomized to receive either study drug or placebo (1.5% NaCl) by inhalation via a PARI eFlow nebulizer. Each subject will complete 28 days of daily dosing. All study patients will be followed for safety, pharmacokinetics, clinical and microbiologic activity for 56 days post completion of study treatment. For the two lower doses (70 mg and 140 mg): patients received drug for 28 days, followed by a 28 day safety evaluation. For 560 mg: patients received drug for 28 days, followed by a 56 day safety evaluation. The total study period will be up to 84 days, with screening visit occurring within the preceding 14 days prior to study day 1. Patients will be clinically evaluated during the first 48 hours post first study dose and weekly for the 28 day treatment period and during the follow up visits at study days 35, 42, 49, 56, 70 and 85 days to determine safety and tolerability, pharmacokinetics (PK) and clinical and microbiologic activity.

Clinical laboratory parameters, audiology testing, clinical adverse events and pulmonary function will be evaluated for all study subjects in order to determine the qualitative and quantitative safety and tolerability of Arikayce™ compared to placebo. Serum, urine and sputum specimens will be collected at periodic intervals to assess PK. Additionally, sputum samples will be collected to determine changes in bacterial density. Pulmonary function testing and CFQ-R measurements will be assessed at selected time points throughout the study. An exploratory evaluation of a Cystic Fibrosis Symptom Diary (CFSD) will also be implemented. Arikace™,Arikayce™, Liposomal Amikacin for Inhalation (LAI), and Amikacin Liposome Inhalation Suspension (ALIS) may be used interchangeably throughout this study and other studies evaluating amikacin liposomal inhalation suspension.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female study subjects must be adults (≥ 6 years of age)
* Confirmed diagnosis of CF
* History of chronic infection with P.aeruginosa
* FEV1 ≥40% of predicted at Screening
* Ability to comply with study medication use, study visits and procedures
* Ability to produce 0.5 grams of sputum

Key Exclusion Criteria:

* Administration of any investigational drug within 8 weeks to Study Day 1
* Emergency room visit or hospitalization for CF or respiratory-related illness within 4 weeks prior to screening
* History of alcohol, medication or illicit drug abuse within 1 yr. to screening
* History of lung transplantation
* Female of childbearing potential who are not practicing an acceptable method of birth control or who are lactating
* Positive Pregnancy test
* Use of any anti-pseudomonal antibiotics within 28 days prior to Study Day 1
* Initiation of chronic therapy within 28 days prior to Study Day 1
* History of sputum or throat swab culture yielding Burkholderia cepacia within 2 years prior to screening
* History of mycobacterial and/or Aspergillus infection requiring treatment within 2 years prior to screening
* History of biliary cirrhosis with portal hypertension, or splenomegaly

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2008-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gina Eagle, MD, Study Director — Insmed Incorporated
Locations (19):
- United States (19):
  - Birmingham, Alabama
  - Los Angeles, California
  - Miami, Florida
  - Orlando, Florida
  - Indianapolis, Indiana
  - Iowa City, Iowa
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Minneapolis, Minnesota
  - Jackson, Mississippi
  - St Louis, Missouri
  - Morristown, New Jersey
  - New Brunswick, New Jersey
  - Albuquerque, New Mexico
  - Rochester, New York
  - Philadelphia, Pennsylvania
  - Sioux Falls, South Dakota
  - Seattle, Washington

REFERENCES:
- [Background] Okusanya OO, Bhavnani SM, Hammel JP, Forrest A, Bulik CC, Ambrose PG, Gupta R. Evaluation of the pharmacokinetics and pharmacodynamics of liposomal amikacin for inhalation in cystic fibrosis patients with chronic pseudomonal infections using data from two phase 2 clinical studies. Antimicrob Agents Chemother. 2014 Sep;58(9):5005-15. doi: 10.1128/AAC.02421-13. Epub 2014 Mar 31. PMID 24687506
- [Derived] Clancy JP, Dupont L, Konstan MW, Billings J, Fustik S, Goss CH, Lymp J, Minic P, Quittner AL, Rubenstein RC, Young KR, Saiman L, Burns JL, Govan JR, Ramsey B, Gupta R; Arikace Study Group. Phase II studies of nebulised Arikace in CF patients with Pseudomonas aeruginosa infection. Thorax. 2013 Sep;68(9):818-25. doi: 10.1136/thoraxjnl-2012-202230. Epub 2013 Jun 8. PMID 23749840
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/24687506

RESULTS

PARTICIPANT FLOW:
Groups:
- Arikayce™ at 560 mg: Subjects randomized 2:1 to receive Arikayce 560 mg or Placebo.
- Placebo at 560 mg: Matching placebo
  Subjects randomized 2:1 to receive Arikayce 560 mg or Placebo.
- Arikayce™ at 70 mg; Arikayce™ at 140 mg: Subjects randomized 1:1:1 to receive Arikayce 70 mg, Arikayce 140 mg or Placebo.
- Placebo at 70mg/140 mg: Matching placebo
  Subjects randomized 1:1:1 to receive Arikayce 70 mg, Arikayce 140 mg or Placebo.
Period: Overall Study
Arm/Group | Arikayce™ at 560 mg | Placebo at 560 mg | Arikayce™ at 70 mg | Arikayce™ at 140 mg | Placebo at 70mg/140 mg
Started | 15 | 7 | 7 | 5 | 7
Completed (completed follow up off treatment) | 12 | 7 | 6 | 5 | 6
Not Completed | 3 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo at 560 mg: Subjects randomized 2:1 to receive Arikayce 560 mg or Placebo.
- Placebo at 70 mg/140 mg: Subjects randomized 1:1:1 to receive Arikayce 70 mg, Arikayce 140 mg or Placebo.
- Total: Total of all reporting groups
Arm/Group | Arikayce™ at 560 mg | Placebo at 560 mg | Arikayce™ at 70 mg | Arikayce™ at 140 mg | Placebo at 70 mg/140 mg | Total
Number analyzed (Participants) | 15 | 7 | 7 | 5 | 7 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Analyses were performed using the modified intent-to-treat (mITT) population, defined as all randomized subjects who received at least one dose of study drug
  years | 31.5 (14.5) | 26.3 (6.7) | 33.1 (9.7) | 35.4 (6.0) | 24.4 (6.3) | 29.9 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Analyses were performed using the modified intent-to-treat (mITT) population, defined as all randomized subjects who received at least one dose of study drug
  Participants
    Female | 5 | 3 | 6 | 1 | 5 | 20
    Male | 10 | 4 | 1 | 4 | 2 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Analyses were performed using the modified intent-to-treat (mITT) population, defined as all randomized subjects who received at least one dose of study drug
  Participants
    White | 14 | 6 | 7 | 5 | 6 | 38
    Black | 1 | 1 | 0 | 0 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 7 | 7 | 5 | 7 | 41

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events
Description: To evaluate the safety and tolerability of 28 days of daily dosing of nebulized Arikayce™, liposomal amikacin for inhalation.
Time Frame: 56 days
Population: Analyses were performed using the modified intent-to-treat (mITT) population, defined as all randomized subjects who received at least one dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Arikayce™ at 560 mg | Placebo at 560 mg | Arikayce™ at 70 mg | Arikayce™ at 140 mg | Placebo at 70mg/140 mg
Number analyzed (Participants) | 15 | 7 | 7 | 5 | 7
Participants
  Patients with AEs | 14 | 7 | 7 | 4 | 6
  Patients with Treatment Related AEs | 7 | 2 | 2 | 2 | 2
  Deaths | 0 | 0 | 0 | 0 | 0
  Patients with Serious AEs | 5 | 2 | 0 | 1 | 1
  Patients Permanently Discontinuing due to AEs | 4 | 0 | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics of Arikayce™ in Serum
Description: Measure PK parameter (Cmax) of Arikayce in serum
Time Frame: Day 1, Day 14 and Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Arikayce™ at 560 mg | Placebo at 560 mg | Arikayce™ at 70 mg | Arikayce™ at 140 mg | Placebo at 70mg/140 mg
Number analyzed (Participants) | 15 | 7 | 7 | 5 | 7
mg/L
  Day 1: number analyzed (Participants) | 15 | 0 | 5 | 5 | 0
  Day 1 | 1.59 (0.973) |  | 0.216 (0.054) | 0.375 (0.167) |
  Day 14: number analyzed (Participants) | 11 | 0 | 7 | 5 | 0
  Day 14 | 2.17 (1.48) |  | 0.265 (0.060) | 0.447 (0.157) |
  Day 28: number analyzed (Participants) | 9 | 0 | 4 | 5 | 0
  Day 28 | 2.71 (1.75) |  | 0.293 (0.026) | 0.481 (0.213) |

3. Secondary Outcome: Pharmacokinetics (PK) of Arikayce™ in Sputum
Description: Measure PK parameters (sputum concentration) of Arikayce in sputum, pre- and post-dose
Time Frame: Day 1 post-dose, Day 14 pre- and post-dose, Day 28 pre- and post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mcg/g
Groups:
- Arikayce ™at 140 mg: Subjects randomized 1:1:1 to receive Arikayce 70 mg, Arikayce 140 mg or Placebo.
Arm/Group | Arikayce™ at 560 mg | Placebo at 560 mg | Arikayce™ at 70 mg | Arikayce ™at 140 mg | Placebo at 70mg/140 mg
Number analyzed (Participants) | 15 | 7 | 7 | 5 | 7
mcg/g
  Day 1 1 hour post-dose: number analyzed (Participants) | 15 | 0 | 7 | 5 | 0
  Day 1 1 hour post-dose | 4417 (74.5) |  | 1119 (64.5) | 1632 (36.9) |
  Day 14 pre-dose: number analyzed (Participants) | 15 | 0 | 7 | 5 | 0
  Day 14 pre-dose | 132 (205) |  | 150 (221) | 20.1 (43.8) |
  Day 14 1 hour post-dose: number analyzed (Participants) | 15 | 0 | 7 | 5 | 0
  Day 14 1 hour post-dose | 2643 (101) |  | 1012 (119) | 1534 (63.3) |
  Day 28 pre-dose: number analyzed (Participants) | 15 | 0 | 7 | 5 | 0
  Day 28 pre-dose | 124 (114) |  | 49.7 (189) | 20.5 (57.0) |
  Day 28 1 hour post-dose: number analyzed (Participants) | 15 | 0 | 7 | 5 | 0
  Day 28 1 hour post-dose | 2670 (66.2) |  | 753 (82.2) | 1468 (90.9) |

4. Secondary Outcome: Pharmacokinetics (PK) of Arikayce™ in Urine
Description: Measure PK parameter (Ae0-24) of Arikayce in urine
Time Frame: Day 1, Day 14 and Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Arikayce™ at 560 mg | Placebo at 560 mg | Arikayce™ at 70 mg | Arikayce ™at 140 mg | Placebo at 70mg/140 mg
Number analyzed (Participants) | 15 | 7 | 7 | 5 | 7
mg
  Day 1: number analyzed (Participants) | 15 | 0 | 6 | 5 | 0
  Day 1 | 25.9 (27.1) |  | 4.80 (1.43) | 15.2 (8.74) |
  Day 14: number analyzed (Participants) | 10 | 0 | 7 | 5 | 0
  Day 14 | 63.6 (29.1) |  | 7.76 (3.19) | 21.7 (12.4) |
  Day 28: number analyzed (Participants) | 9 | 0 | 6 | 5 | 0
  Day 28 | 62.9 (38.0) |  | 7.13 (4.31) | 17.7 (8.33) |

5. Secondary Outcome: Pharmacokinetics (PK) of Arikayce™ in Serum
Description: Measure PK parameter (AUC) of Arikayce in Serum
Time Frame: Day 1, Day 14 and Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg*hr/L
Arm/Group | Arikayce™ at 560 mg | Placebo at 560 mg | Arikayce™ at 70 mg | Arikayce ™at 140 mg | Placebo at 70mg/140 mg
Number analyzed (Participants) | 15 | 7 | 7 | 5 | 7
mg*hr/L
  Day 1: number analyzed (Participants) | 15 | 0 | 7 | 5 | 0
  Day 1 | 11.3 (5.81) |  | 1.06 (0.243) | 2.90 (1.08) |
  Day 14: number analyzed (Participants) | 15 | 0 | 7 | 5 | 0
  Day 14 | 15.0 (7.96) |  | 1.56 (0.553) | 4.32 (1.96) |
  Day 28: number analyzed (Participants) | 15 | 0 | 7 | 5 | 0
  Day 28 | 17.1 (7.58) |  | 1.59 (0.531) | 4.16 (1.56) |

6. Secondary Outcome: Pulmonary Function: Pre-Dose FEV1 (%-Predicted)
Description: Relative Change (%) from Baseline to Day 28, Day 56, Day 70, and Day 84 in Pulmonary Function
Time Frame: Baseline, Day 28, Day 56, Day 70 and Day 84
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent (%)
Arm/Group | Arikayce™ at 560 mg | Placebo at 560 mg | Arikayce™ at 70 mg | Arikayce™ at 140 mg | Placebo at 70mg/140 mg
Number analyzed (Participants) | 15 | 7 | 7 | 5 | 7
Percent (%)
  Baseline | 68.800 (17.026) | 66.143 (12.020) | 59.286 (12.593) | 70.400 (10.090) | 69.286 (16.550)
  Day 28: number analyzed (Participants) | 13 | 7 | 7 | 5 | 7
  Day 28 | -0.003 (0.124) | -0.001 (0.075) | 0.029 (0.124) | -0.029 (0.089) | -0.010 (0.060)
  Day 56: number analyzed (Participants) | 13 | 7 | 7 | 5 | 6
  Day 56 | 0.029 (0.092) | -0.028 (0.129) | 0.024 (0.076) | -0.020 (0.087) | 0.011 (0.067)
  Day 70: number analyzed (Participants) | 12 | 7 | 0 | 0 | 0
  Day 70 | 0.026 (0.107) | -0.043 (0.097) |  |  |
  Day 84: number analyzed (Participants) | 12 | 7 | 0 | 0 | 0
  Day 84 | 0.000 (0.078) | -0.067 (0.145) |  |  |

7. Secondary Outcome: Density of Pseudomonas Aeruginosa in Sputum
Description: Change (log10 CFU) from Baseline by Study Day and Treatment Arm
Time Frame: Day 7, Day 14, Day 21, Day 28 and Day 35
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Log 10 CFU/g
Arm/Group | Arikayce™ at 560 mg | Placebo at 560 mg | Arikayce™ at 70 mg | Arikayce™ at 140 mg | Placebo at 70mg/140 mg
Number analyzed (Participants) | 15 | 7 | 7 | 5 | 7
Log 10 CFU/g
  Day 7: number analyzed (Participants) | 13 | 5 | 7 | 5 | 5
  Day 7 | -1.605 (1.308) | 1.118 (2.214) | -1.093 (0.616) | -0.637 (0.711) | -0.254 (0.991)
  Day 14: number analyzed (Participants) | 10 | 5 | 6 | 5 | 5
  Day 14 | -1.082 (1.354) | 1.098 (2.477) | -1.121 (1.404) | -0.175 (1.014) | -0.159 (0.499)
  Day 21: number analyzed (Participants) | 10 | 5 | 6 | 5 | 4
  Day 21 | -0.750 (1.466) | -0.057 (0.600) | -1.560 (2.845) | -0.255 (1.977) | -0.337 (1.384)
  Day 28: number analyzed (Participants) | 11 | 4 | 6 | 5 | 3
  Day 28 | -1.576 (1.979) | 0.836 (1.544) | -1.771 (1.741) | -0.381 (0.660) | -0.426 (0.435)
  Day 35: number analyzed (Participants) | 10 | 4 | 4 | 5 | 4
  Day 35 | -1.963 (2.456) | 0.578 (0.539) | -0.675 (0.452) | 0.256 (1.058) | 0.028 (0.243)

8. Secondary Outcome: Duration of Systemic Anti-Pseudomonal Rescue Therapy
Time Frame: Through study duration, approximately 84 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Arikayce™ at 560 mg | Placebo at 560 mg | Arikayce™ at 70 mg | Arikayce™ at 140 mg | Placebo at 70mg/140 mg
Number analyzed (Participants) | 15 | 7 | 7 | 5 | 7
days | 22.800 (12.778) | 30.333 (15.044) | 17.500 (4.950) | 18.000 (0) | 30.500 (10.607)

9. Secondary Outcome: CFQ-R Respiratory Scale (Relative Change % From Baseline)
Description: Quality of Life was measured by the absolute change from baseline in the Cystic Fibrosis Questionnaire-Revised (CFQ-R) respiratory scale. Disease specific instrument designed to measure impact on overall health, daily life, perceived well-being and symptoms in patients with a diagnosis of cystic fibrosis. Scores range from 0 to 100, with higher scores indicating better health. Scores for each Health Related Quality of Life (HRQoL) domain; after recoding, each item is summed to generate a domain score and standardized.
Time Frame: Day 15, Day 28 and Day 42
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent (%)
Arm/Group | Arikayce™ at 560 mg | Placebo at 560 mg | Arikayce™ at 70 mg | Arikayce ™at 140 mg | Placebo at 70mg/140 mg
Number analyzed (Participants) | 15 | 7 | 7 | 5 | 7
Percent (%)
  Day 15: number analyzed (Participants) | 13 | 7 | 7 | 5 | 7
  Day 15 | 0.385 (0.638) | -0.063 (0.135) | 0.075 (0.273) | 0.100 (0.173) | 0.042 (0.104)
  Day 28: number analyzed (Participants) | 12 | 7 | 6 | 4 | 7
  Day 28 | 0.387 (0.683) | -0.054 (0.229) | 0.126 (0.255) | 0.228 (0.304) | -0.029 (0.233)
  Day 42: number analyzed (Participants) | 10 | 6 | 5 | 4 | 7
  Day 42 | 0.094 (0.826) | -0.084 (0.258) | -0.012 (0.305) | 0.225 (0.215) | 0.006 (0.173)

ADVERSE EVENTS:
Groups:
- Placebo at 70 mg/140 mg: Matching placebo
  Subjects randomized 1:1:1 to receive Arikayce 70 mg, Arikayce 140 mg or Placebo.
Arm/Group | Arikayce™ at 560 mg | Placebo at 560 mg | Arikayce™ at 70 mg | Arikayce™ at 140 mg | Placebo at 70 mg/140 mg
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/7 | 0/7 | 0/5 | 0/7
Serious Adverse Events (participants affected / at risk) | 5/15 | 2/7 | 0/7 | 1/5 | 1/7
Other Adverse Events (participants affected / at risk) | 14/15 | 7/7 | 7/7 | 4/5 | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arikayce™ at 560 mg (N=15) | Placebo at 560 mg (N=7) | Arikayce™ at 70 mg (N=7) | Arikayce™ at 140 mg (N=5) | Placebo at 70 mg/140 mg (N=7)
LOBE PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary exacerbation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cystic Fibrosis Exacerbation (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
migraine headaches (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Elevated LFTs (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arikayce™ at 560 mg (N=15) | Placebo at 560 mg (N=7) | Arikayce™ at 70 mg (N=7) | Arikayce™ at 140 mg (N=5) | Placebo at 70 mg/140 mg (N=7)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 | 0 | 1
Chills (General disorders) | 2 (2) | 0 (0) | 0 | 1 | 1
Fatigue (General disorders) | 2 (2) | 0 (0) | 2 | 1 | 1
Non cardiac chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 1 (1) | 0 | 0 | 2
ALT increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
AST increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Migraine (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3) | 1 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea, exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 | 1 | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 | 1 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 1 (1) | 2 | 1 | 3
Nasal edema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 2 | 1 | 1
Prolonged expiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 | 1 | 1
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Throat Tightness (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 2 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2
Vessel Puncture site hematoma (General disorders) | 0 (0) | 0 (0) | 1 | 0 | 1
Creatinine Renal Clearance INcreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 | 1 | 1
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Per the signed Investigator Agreement in the study protocol and protocol amendments, the PI agreed "not to originate or use the name of Insmed Incorporated, or study drug code in any publicity, news release, or other public announcement, written or oral, whether to the public, press, or otherwise, relating to this protocol, to any amendment to the protocol, or to the performance of this protocol, without the prior written consent of Insmed Incorporated."